CLINICAL TRIAL: NCT06460688
Title: Effects Of Mother Rehabilitative Aid Education Program On Parental Stress And Gross Motor Function Among Children With Diplegic Cerebral Palsy
Brief Title: Effect of Mother Rehabilitative Aid Education Program on Children With Diplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/07102
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Diplegic Cerebral Palsy
Keywords: Cerebral Palsy; Gross Motor Function; Mother Rehabilitative Aid; Parental Stress; Spastic Diplegic
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: It will be Randomized control trial in which non probability convenient sampling will be used. two groups of age 6-12will be formed in which participants will be randomly divided. Group A will receive Mother Rehabilitative Aid Education program with routine neurophysical therapy and Group B will only receive routine neurophysical therapy
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mother Rehabilitative Aid Education Program (Experimental): Participants in group A will be educate thoroughly about treatment plan which includes routine neuro physical therapy aiming (Gross Motor Function & Balance) A class will be organized to educate Mothers/ Caregivers through PPT presentation, video and pictures. This class will contain 3 domains (Counseling, Educating, Practicing). Feedback will be taken on daily basis through video recordings. Mothers will take part in treatment session, 45 minutes for 5 days a week for 8 weeks.
  Interventions: Other: Mother Rehabilitative Aid Education Program
- Neuro physical Therapy. (Active Comparator): Routine neuro physical therapy will be given(1) for 45 minutes, 5 days a week for 8 weeks. Participants in group B will not be educated about treatment plan. Routine home plan was given in this group once in a week, for 8 weeks.
  Interventions: Other: Neuro physical Therapy

INTERVENTIONS:
Other: Mother Rehabilitative Aid Education Program — Routine neuro physical therapy will be given which includes Stretching, truck control and independent transition, train standing and activation of base, gain walking with minimal assistance, Gain ground clearance with stair climbing. A class will be organized to educate Mothers/ Caregivers through PPT presentation, video and pictures. This class will contain 3 domains (Counseling, Educating, Practicing). Feedback will be taken on daily basis through video recordings. Mothers will take part in treatment session, 45 minutes for 5 days a week for 8 weeks.
  Arms: Mother Rehabilitative Aid Education Program
Other: Neuro physical Therapy — Routine neuro physical therapy will be given which includes Stretching, truck control and independent transition, train standing and activation of base, gain walking with minimal assistance, Gain ground clearance with stair climbing. for 45 minutes, 5 days a week for 8 weeks. Participants in group B will not be educated about treatment plan. Routine home plan was given in this group once in a week, for 8 weeks.
  Arms: Neuro physical Therapy.

SUMMARY:
Cerebral palsy (CP) is a syndrome caused by a non-progressive lesion in the developing brain. Spastic diplegia cerebral palsy is a form of cerebral palsy, permanently affects muscle control and coordination. Symptoms include increased muscle tone which leads to spasticity (stiff or tight muscles and exaggerated reflexes) in the legs. Physiotherapist will come across many children with disability and it's a daily routine that providing treatment and educating parents regarding the treatment and ask them to continue at home. Family centered home program for children with disability plays a major role in their improvement. By educating and creating awareness among mother's, it can really do justice for the recovery of differently abled children.

This will be a randomized control trial. Study will be conducted on 24 patients. Inclusion criteria of this study is mothers of spastic cerebral palsy children (Diplegic), Age 6-12 years, with GMFCS level II & III and mothers who are willing to spend time in giving home program and give feedback every day and should maintain continuity coming to the department. Mothers of Cerebral palsy (diplegic) children will be excluded if the children are suffering with fixed deformities and with recent surgeries involving spine and limbs. Working females more than 5 working hours are also excluded. Participants will be divided randomly into two groups. In group A, Participants will be educated thoroughly about treatment plan which includes routine neuro physical therapy aiming (Gross Motor Function & Balance). A class will be organized to educate Mothers/ Caregivers through PPT presentation, video and pictures. In group B, participants will not be educated about treatment plan, routine home plan was given once in a week. Intervention will be given for 8 weeks, 5 days a week for 45 minutes. Pre and post session Gross motor function by GMFM, balance by PBS, Quality of life by CP-QOL and parental stress by PSI will be measured.

DETAILED DESCRIPTION:
Participants in group A will be educate thoroughly about treatment plan which includes routine neuro physical therapy aiming (Gross Motor Function & Balance)which includes (To reduce the spasticity of the muscle by sustained passive stretching of hamstring, tendo-achilles, and adductors (30 secs hold * 3 rep), once a day, five times a week for 8 weeks, Gain trunk control and independent transition by sit to stand facilitation on bolster (5 rep), progressing with single leg sit to stand (5 rep) and multidirectional reach-outs in sitting for five times a week for 8 weeks, train standing and activation of base, Standing training, in which the child was asked to stand while receiving maximum support at the pelvis and knees. After two or more weeks, we began assisting them in taking a few steps with minimal pelvic support. Task oriented approaches were added to facilitate weight shifting for five times a week for 8 weeks, Gain walking with minimal assistance by Gait training with minimal pelvic support assistance. Stepping forward and reach outs for five times a week for 8 weeks. Gain ground clearance and stair climbing by step up and step-down facilitation with stepper and progressing with doing on stair case for 5 times a week for 8 weeks). A class will be organized to educate Mothers/ Caregivers through PPT presentation, video and pictures. This class will contain 3 domains (Counseling, Educating, Practicing). Feedback will be taken on daily basis through video recordings. Mothers will take part in treatment session, 45 minutes for 5 days a week for 8 weeks. In Group B Routine neuro physical therapy will be given for 45 minutes, 5 days a week for 8 weeks. Participants in group B will not be educated about treatment plan. Routine home plan was given in this group once in a week, for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of spastic cerebral palsy children (Diplegic)
* Mothers of children spastic diplegic CP age 6-12 years either gender
* Mothers of children spastic diplegic CP with GMFCS level II & III
* Mothers who are willing to spend time in giving home program and give a feedback every day and should maintain continuity coming to the department.

Exclusion Criteria:

* Mothers of Cerebral palsy children will be excluded if the children are suffering with fixed deformities.
* Mothers of children having spastic CP with recent surgeries involving spine and limbs
* Working females (>5 hours working time)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-07-21 (Actual); Study Completion 2024-07-28 (Actual)

PRIMARY OUTCOMES:
GMFM-88 (Gross Motor Function Measure) | 8 weeks
  The Gross Motor Function Measure (GMFM) is a tool that has been developed to assess change in gross motor function in children with cerebral palsy aged 5 months to 16 years of age. The 88 items are grouped into five dimensions: 1) lying and rolling, 2) sitting, 3) crawling and kneeling, 4) standing, and 5) walking, running and jumping. A maximum of three trials is allowed for each item and the best trial is recorded. Scores for each dimension are expressed as a percentage of the maximum score for that dimension and the total score is obtained by averaging the percentage scores across the five dimensions.
Parental Stress Index | 8 weeks
  The degree of parental stress was evaluated with the Parenting Stress Index (PSI) (Abidin and Wilfong 1989). The PSI is designed to identify stressful areas in parent child interactions, and the results from the PSI indicate whether parents experience distress to a clinically disturbing degree. The Parenting Stress Index Short Form was standardized for use with parents of children ranging from 1 month to 12 years old.

SECONDARY OUTCOMES:
CP-QOL ( Quality of life) | 8 weeks
  The CP QOL-Child was designed to assess several aspects of subjective happiness and well-being, rather than ill-being or functioning. It is useful to establish a profile of qualify of life of children with CP to understand their subjective perception of their life (Waters et al., 2009, Waters et al., 2005). Two versions of the CP QOL-Child are available: a primary caregiver-proxy report version (proxy version) for children aged 4-12 years (which we are using), and a self-report version for children aged 9-12 years. The reliability and validity of the CP QOL-Child have been established, including internal consistency, test-retest reliability, and construct validity (Wang et al., 2010, Waters et al., 2007)(19)

CONTACTS AND LOCATIONS:
Overall Officials: Izza Akmal, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah Internationl University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harjpal P, Raipure A, Kovela RK, Qureshi MI. The Effect of Neuro-Physiotherapy on Gross Motor Function in a Male Child With Spastic Diplegic Cerebral Palsy: A Case Report. Cureus. 2022 Sep 19;14(9):e29310. doi: 10.7759/cureus.29310. eCollection 2022 Sep. PMID 36277570